CLINICAL TRIAL: NCT07047937
Title: Explainable Machine Learning for Predicting Early Gastric Cancer: a Retrospective Cohort Study
Brief Title: Explainable Machine Learning for Predicting Early Gastric Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Wenzhou Central Hospital (Other)
Responsible Party: Principal Investigator, sunmeng chen, Resident in gastrointestinal surgery, Wenzhou Central Hospital
Other Study IDs: 202506031607000064611
Record Dates: First submitted 2025-06-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Early Gastric Cancer
Keywords: early detection of cancer; early gastric cancer; machine learning; prediction model; SHapley Additive exPlanation (SHAP)
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abstract Background: Early detection of gastric cancer is crucial for improving patient survival rates. Currently, the primary method for diagnosing early-stage gastric cancer is endoscopy, which has various limitations. Additionally, single laboratory tests continue to fall short of the requirements for early screening. This study aims to develop a machine learning (ML) model using clinical data to predict early-stage gastric cancer and apply SHapley Additive exPlanation (SHAP) values to explain the ML model.

Methods: This study involved patients who provided gastric tissue samples at Wenzhou Central Hospital from 2019 to 2023. The investigators gathered various laboratory test results from these patients. The investigators constructed and evaluated nine ML models to predict early-stage gastric cancer, using the area under the curve (AUC), accuracy, and sensitivity to assess their performance. For the most effective prediction model, The investigators utilized the SHAP method to determine the features' importance and explain the ML model.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a gastric tissue pathology result are included

Exclusion Criteria:

* unclear or incomplete pathology results
* significant missing laboratory data
* progressive and advanced gastric cancer

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients with a gastric tissue pathology result are included,1,085 patients were included in the study
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Explainable machine learning for predicting early gastric cancer | From June 2025 to July 2025
  The area under the ROC curve (AUC) was used as the primary outcome measure

SECONDARY OUTCOMES:
Explainable machine learning for predicting early gastric cancer | From June 2025 to July 2025
  We considered the sensitivity of the model as a secondary outcome measure.

OTHER OUTCOMES:
Explainable machine learning for predicting early gastric cancer | From June 2025 to July 2025
  We included model accuracy as other outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenzhou Central Hospital, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial.
Supporting Information: Study Protocol
Time Frame: Approximately from August 1, 2025 to November 1, 2025.
Access Criteria: Log in to the clinical trial public management platform, and researchers can query the original research records and data of the research plan on this platform.
URL: http://www.medresman.org.cn